CLINICAL TRIAL: NCT06647550
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Dose-finding, Phase 2 Study to Assess the Efficacy and Safety of HD-6277 in Adult Patients With Inadequate Control of Type 2 Diabetes Mellitus by Diet and Exercise
Brief Title: To Assess the Efficacy and Safety of HD-6277 in Adult Patients With Inadequate Control of Type 2 Diabetes Mellitus by Diet and Exercise
Acronym: HDNO-1605
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hyundai Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HT-006-04
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HD-6277 100mg tab (Experimental): Oral tablet
  Interventions: Drug: HD-6277 100mg
- HD-6277 50mg tab (Experimental): Oral tablet
  Interventions: Drug: HD-6277 50mg
- HD-6277 25mg tab (Experimental): Oral tablet
  Interventions: Drug: HD-6277 25mg
- Placebo (Placebo Comparator): Oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HD-6277 100mg — PO, QD
  Arms: HD-6277 100mg tab
Drug: HD-6277 50mg — PO, QD
  Arms: HD-6277 50mg tab
Drug: HD-6277 25mg — PO, QD
  Arms: HD-6277 25mg tab
Drug: Placebo — PO, QD
  Arms: Placebo

SUMMARY:
A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Dose-finding, Phase 2 Study to Assess the Efficacy and Safety of HD-6277 in Adult Patients with Inadequate Control of Type 2 Diabetes Mellitus by Diet and Exercise

DETAILED DESCRIPTION:
This trial is a phase 2 study to evaluate the efficacy and safety of HD-6277 in Adult Patients with Inadequate Control of Type 2 Diabetes Mellitus by Diet and Exercise.

This is multi-center, double-blind, placebo-controlled, parallel-group, dose-finding phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM with HbA1c between 7.0% and 10.0% (inclusive) while on diet and exercise alone for at least 8 weeks prior to screening.

Exclusion Criteria:

* Type 1 diabetes or another immune-mediated diabetes syndrome
* BMI: > 40 kg/m2
* C-peptide: < 0.5ng/mL

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
change in HbA1c at weeks 12 from baseline | at weeks 12 from baseline
  change in HbA1c at weeks 12 from baseline

SECONDARY OUTCOMES:
change in HbA1c at weeks 6 from baseline | at weeks 6 from baseline
  change in HbA1c at weeks 6 from baseline
percentage of subjects with HbA1c level below 7.0% at weeks 12 | at weeks 12
  percentage of subjects with HbA1c level below 7.0% at weeks 12
percentage of subjects with HbA1c level below 6.5% at weeks 12 | at weeks 12
  percentage of subjects with HbA1c level below 6.5% at weeks 12
change in Glycoalbumin at weeks 6 and 12 from baseline | at weeks 6 and 12 from baseline
  change in Glycoalbumin at weeks 6 and 12 from baseline

OTHER OUTCOMES:
change in body weight at weeks 6 and 12 from baseline | at weeks 6 and 12 from baseline
  change in body weight at weeks 6 and 12 from baseline
change in GA/HbA1c at weeks 6 and 12 from baseline | at weeks 6 and 12 from baseline
  change in GA/HbA1c at weeks 6 and 12 from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No